CLINICAL TRIAL: NCT05432869
Title: Effects of External Electrical Stimulating Applied on the Thigh in Men With Urinary Incontinence After Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/06/22
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical stimulation (ES) group (Experimental): ES group will be given additional external electrical stimulation to the lifestyle advices.
  Interventions: Other: ES and lifestyle advices
- Control group (Experimental): Control group will be given only lifestyle advices .
  Interventions: Other: Lifestyle advices

INTERVENTIONS:
Other: ES and lifestyle advices — The lifestyle advices include fluid consumption, diet, weight control, constipation, smoking, etc.
  External electrical stimulation will be applied for 30 minutes 3 days a week during 4 weeks. Electrodes were placed on the thighs.
  Arms: Electrical stimulation (ES) group
Other: Lifestyle advices — The lifestyle advices include fluid consumption, diet, weight control, constipation, smoking, etc.
  Arms: Control group

SUMMARY:
The aim of this study is to investigate the effects of external electrical stimulation applied on the thigh on urinary symptoms, quality of life, sexual function, perception of subjective improvement and satisfaction in men with urinary incontinence after prostatectomy

DETAILED DESCRIPTION:
The most common complication after prostatectomy surgeries is urinary incontinence. There are conservative and surgical treatment options in post-prostatectomy urinary incontinence. One of the conservative treatment options is electrical stimulation application.

Electrical stimulation with the intraanal probe in men is painful and uncomfortable.

And also there are few studies, demonstrating the effects of electrical stimulation on urinary incontinence after prostatectomy in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being a male individual with stress or stress-dominant mixed urinary incontinence symptoms after undergoing prostatectomy surgery
* Being over 40 years old
* Not having residual cancerous tissue
* Volunteering to participate in the study

Exclusion Criteria:

* Having serious cardiovascular disease (unstable angina and arrhythmia patients, heart failure patients, etc.)
* Having sensory loss
* Having an ongoing urinary infection
* Having only urgency urinary incontinence
* Using a pacemaker
* Receiving active cancer treatment (radiotherapy, chemotherapy)
* Those who have a problem that interferes with cooperation and understanding

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with urinary incontinence after prostatectomy
Enrollment: 40 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence severity | change from baseline at 4 weeks
  Urinary incontinence severity will be assessed with a 1-hour pad test. This amount; less than 2 grams is considered normal, 2-10 grams is mild, 10-50 grams is moderate, and over 50 grams is severe stress urinary incontinence.

SECONDARY OUTCOMES:
Presence of urinary incontinence symptoms | change from baseline at 4 weeks
  Urinary incontinence symptoms will be assessed with International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF). It consists of 6 questions in total and the total score is 3., 4., 5. It is obtained by adding the scores they get from the questions. A low score in the scale indicates that urinary incontinence symptoms are less.
Life quality | change from baseline at 4 weeks
  Life quality will be assessed with King Health Questionnaire. The questionnaire, consisting of thirty-two items, consists of 2 parts. In the first part, there are 2 questions questioning the general health perception and incontinence effect, and 19 questions dividing the quality of life into 7 areas (role limitations, physical limitations, social limitations, personal relationships, emotional problems, sleep/energy disorders, symptom severity measurement). In the second part, there are 11-item complaint severity scales that evaluate the presence and severity of urinary symptoms. While the best score that can be obtained on the complaint severity scale is "0", the worst score is "30", the best score that can be obtained for all King Health Questionnaire subsections is "0" and the worst score is "100".
Sexual function | change from baseline at 4 weeks
  Sexual function will be assessed with International Index of Erectile Function-5. It includes 5 main topics; erectile function, orgasm function, sexual desire, sexual intercourse satisfaction and general satisfaction are questioned with a total of 5 questions. Each question gets a score between 0-5. Total score; severe (5-7), moderate (8-11), mild-moderate (12-16), mild (17-21), no erectile dysfunction (22-25)
Perception of Subjective Improvement | after treatment (4th week)
  Patients' subjective perception of improvement will be questioned with a 4-point Likert scale (worse (1), same (2), better (3) and completely cured (4))
Patients Satisfaction | after treatment (4th week)
  Patient satisfaction will be questioned with a 5-point Likert scale (not at all satisfied (1), dissatisfied (2), undecided (3), satisfied (4), very satisfied (5))
Compliance with Lifestyle Advices | after treatment (4th week)
  Compliance of patients to the lifestyle advices will be evaluated using a 100-mm visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University